CLINICAL TRIAL: NCT04079348
Title: Feasibility Study to Compare OASIS Extracellular Matrix to Standard Wound Care for Treatment of Donor Site Wounds
Brief Title: Oasis Donor Site Wounds Post-Market Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Biotech Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-001
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Surgical Wound; Wound; Wounds and Injuries; Wound Heal
Keywords: Donor Site Wound
MeSH Terms: conditions — Surgical Wound; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: A patient is suitable for inclusion in the study if the patient meets the following criteria, based on known information at the time of enrolment:
  1. Has a split thickness skin graft (STSG) donor site wound no greater than 14 x 20 cm in size requiring placement of a covering material.
Who Masked: Outcomes Assessor
Masking Description: Randomization to treatment groups will be performed using a computer system to randomly assign subjects to treatment arms. Sealed envelopes numbered 1-40 will be provided to the study site. Patients will be assigned an envelope number upon providing informed consent. The envelope will be opened during the treatment procedure to minimize the risk of bias in patient assignment to the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Oasis ECM (Active Comparator): The patient will undergo harvesting of a split-thickness skin graft using a dermatome set at standard depth with the subsequent application Oasis Extracellular Matrix to their donor site wound.
  Interventions: Device: Oasis ECM
- Standard wound care (Active Comparator): The patient will undergo harvesting of a split-thickness skin graft using a dermatome set at standard depth with the subsequent application of standard wound care to their donor site wound.
  Interventions: Other: standard wound care

INTERVENTIONS:
Device: Oasis ECM — The patient will undergo harvesting of a split-thickness skin graft using a dermatome set at standard depth with the subsequent application of Oasis Extracellular Matrix to their donor site wound.
  Arms: Oasis ECM
Other: standard wound care — The patient will undergo harvesting of a split-thickness skin graft using a dermatome set at standard depth with the subsequent application of standard wound care to their donor site wound.
  Arms: Standard wound care

SUMMARY:
The purpose of this study is to demonstrate the safety and performance of Oasis extracellular matrix (ECM) when used as a treatment for donor site wounds in the United Kingdom. Oasis ECM is commercially available for the treatment of partial and full-thickness skin wounds, including chronic wounds, wounds from trauma, and wounds that occur during surgery, such as donor site wounds. The ability of the Oasis ECM to promote the healing of donor site wounds will be evaluated in this study.

About 40 patients (20 in each arm) over 16 years old will be involved in this study at one center in the United Kingdom.

ELIGIBILITY:
Inclusion Criteria:

1. Has a split thickness skin graft (STSG) donor site wound no greater than 14 x 20 cm in size requiring placement of a covering material.
2. Has at least 24 hours to consent to study participation.

Exclusion Criteria:

1. Age < 16 years
2. Patients who, in the opinion of the investigator, have co-morbidities that impair wound healing, such as:

   1. Chronic inflammatory skin condition
   2. Chronic liver failure
   3. Chronic renal failure
   4. Blood-borne viruses (Hep B, Hep C, HIV)
   5. Peripheral vascular disease
   6. Clinically significant anaemia
   7. Uncontrolled diabetes
3. Need for use of the same harvest site (re-cropping)
4. History of radiation therapy to proposed donor site
5. Chronic use of medications known to impair wound healing
6. Chronic use of opioids or neuropathic pain agents
7. Suspected cellulitis, osteomyelitis or septicaemia
8. Patients undergoing haemodialysis
9. Patients requiring spinal/regional block
10. Patients on current anti-coagulant therapy
11. Unable or unwilling to provide informed consent
12. Unable or unwilling to comply with the study follow-up schedule, and procedures
13. Simultaneously participating in another investigational drug or device study (patient must have completed the follow-up phase for the primary endpoint of any previous study at least 30 days prior to enrolment in this study)
14. Allergy or hypersensitivity to materials that are porcine-based
15. Cultural or religious objection to the use of pig or porcine products
16. Known intolerance/allergy to standard wound care products
17. Presence of a local infection at the donor site and/or systemic infection

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Donor site wound healing | 14 days
  To demonstrate the percentage of patients with wounds healed at day 14

SECONDARY OUTCOMES:
Amount of pain, analgesic usage | 14 days
  Patient will record daily usage of analgesics in a diary, daily, over the first 14 days post-treatment
Amount of pain, patient perceived | 14 days
  Patient will use the Visual Analog Score (VAS) to record pain in a diary, daily, over the first 14 days post-treatment.
Cosmetic Outcome utilizing POSAS | up to 6 months
  Cosmesis of the donor site wound will be assessed 3- and 6-months post-treatment by using the Patient and Observer Scar Assessment Scale (POSAS).
Adverse Events | up to 6 months
  Summary of adverse events reported

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No